CLINICAL TRIAL: NCT07204301
Title: Enhancing Patient Comfort and Reducing Anxiety During Flexible Cystoscopy and Bladder Instillation in Bladder Cancer Patients: A Randomized Controlled Trial and Observational Study
Acronym: Flexi-comfort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Nicholas Power, Principle Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16395
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer
Keywords: flexible cystoscopy; bladder instillation; Patient comfort; Anxiety reduction; Pain management; Urologic oncology; Bladder cancer surveillance; Patient-reported outcomes; Procedural anxiety; Minimally invasive urology
MeSH Terms: conditions — Urinary Bladder Neoplasms; Agnosia | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a parallel fashion to either standard care or comfort-enhancing interventions during flexible cystoscopy or intravesical instillation. Each participant will remain in their assigned group for the duration of the study, and outcomes will be compared between groups.
  The interventions include practical, non-pharmacologic strategies (e.g., optimized timing of anesthetic gel, calming music, visual distraction, or ambient lighting changes) that can be readily implemented in routine urologic practice. This design allows assessment of the effectiveness of each intervention compared with usual care in a real-world procedural setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No Intervention (No Intervention): Usual flexible cystoscopy or intravesical instillation under routine clinic conditions. Local anesthetic gel used per usual practice; no added comfort intervention.
- Optimized Anesthetic Gel Timing (Experimental): 2% lidocaine uro-gel instilled before and after procedure to maximize mucosal anesthesia.
  Interventions: Other: Optimized Timing of Intravesical Lidocaine Gel
- Calming Music (Experimental): Patients listen to a standardized calming playlist via headphones during the procedure.
  Interventions: Behavioral: Calming Music During Procedure
- Visual Distraction (Experimental): Patients view standardized visual content on a tablet/monitor positioned for comfort-focused distraction.
  Interventions: Behavioral: Visual Distraction with Screen Content
- Ambient Lighting (Experimental): Procedure performed under standardized calming ambient lighting (blue-hue) per protocol.
  Interventions: Other: Calming Ambient Lighting
- Peak-End Modification (Experimental): At the end of the procedure the flexible cystoscope is deliberately left in the bladder for 2 minutes, without manipulation, to reduce intensity/discomfort, based on the psychological principle of the "peak-end rule," aiming to improve overall remembered experience of the procedure.
  Interventions: Behavioral: Peak-End Modification of Procedure

INTERVENTIONS:
Other: Optimized Timing of Intravesical Lidocaine Gel — Procedural modification of intravesical anesthetic gel administration. Lidocaine gel is instilled before and after flexible cystoscopy or bladder instillation to optimize mucosal anesthesia. This differs from standard practice where timing is not standardized - usually just before flexible cystoscopy.
  Other Names: Anesthetic Gel Timing Modification; Lidocaine Gel Administration Interval
  Arms: Optimized Anesthetic Gel Timing
Behavioral: Calming Music During Procedure — Participants listen to a standardized playlist of calming instrumental music delivered through headphones during the procedure. Intervention is intended to reduce procedural anxiety and discomfort.
  Other Names: Relaxing Music; Music Therapy
  Arms: Calming Music
Behavioral: Visual Distraction with Screen Content — Participants watch standardized visual content (e.g., relaxing video) on a screen or tablet during cystoscopy or bladder instillation. Designed to distract attention and enhance comfort.
  Other Names: Video Distraction; Screen Viewing
  Arms: Visual Distraction
Other: Calming Ambient Lighting — Flexible cystoscopy or intravesical instillation performed under standardized calming ambient lighting (blue-hue) instead of standard clinical lighting. Intervention aims to promote relaxation and reduce anxiety.
  Other Names: Lighting Modification
  Arms: Ambient Lighting
Behavioral: Peak-End Modification of Procedure — Modification of the procedural ending based on the psychological "peak-end rule." The end of the cystoscopy or instillation is deliberately altered to reduce final discomfort, aiming to improve overall remembered patient experience.
  Other Names: Peak-End Rule Adjustment
  Arms: Peak-End Modification

SUMMARY:
The goal of this clinical trial is to learn if certain comfort-enhancing interventions can reduce pain and anxiety during flexible cystoscopy and bladder instillation in patients with bladder cancer. The main questions it aims to answer are:

* Do these interventions reduce patient-reported anxiety during the procedure?
* Do these interventions reduce patient-reported pain or discomfort during the procedure?

Researchers will compare patients receiving comfort interventions (such as timing of anesthetic gel, calming music, or visual distraction) to those receiving standard care to see if these changes improve patient experience.

Participants will:

* Undergo a flexible cystoscopy or bladder instillation as part of their usual care
* Be randomly assigned to receive one or more comfort interventions, or standard care
* Complete short questionnaires about their pain, comfort, and anxiety

DETAILED DESCRIPTION:
Bladder cancer is one of the most common malignancies of the urinary tract, and many patients require frequent endoscopic procedures as part of diagnosis, treatment, and surveillance. Flexible cystoscopy and intravesical instillation are standard procedures but are often associated with patient discomfort, anxiety, and negative procedural experiences. Improving comfort during these procedures has the potential to increase patient satisfaction, reduce procedural avoidance, and improve adherence to follow-up care.

Rationale Although flexible cystoscopy is minimally invasive, it can cause pain, embarrassment, and significant anxiety. Standard strategies to improve patient comfort, such as intravesical anesthetic gel, are variably effective. Previous work suggests that environmental modifications (e.g., calming music, ambient lighting), behavioral strategies (e.g., distraction), and optimization of local anesthetic use may enhance the patient experience. However, rigorous randomized controlled data in the cystoscopy and bladder instillation setting are lacking.

This study will address this gap by systematically evaluating comfort-enhancing interventions during flexible cystoscopy and bladder instillation for bladder cancer patients.

Study Objectives The primary objective is to determine whether comfort interventions reduce patient-reported anxiety and pain during flexible cystoscopy and bladder instillation procedures.

Secondary objectives include:

* To assess whether these interventions improve overall patient satisfaction.
* To determine whether these interventions influence willingness to undergo repeat procedures.
* To explore procedural efficiency, clinician satisfaction, and feasibility of implementing these interventions in routine care.

Study Design This study includes both a randomized controlled trial (RCT) and an observational component.

Randomized Controlled Trial (Interventional Arm):

Participants will be randomly assigned to receive standard care or a comfort interventions, such as:

* Optimized timing of intravesical anesthetic gel
* Calming background music
* Visual distraction or environmental modifications
* Ambient lighting changes

Outcomes will be assessed using validated questionnaires (e.g., visual analogue scales for pain and anxiety, standardized patient-reported outcome measures).

Observational Arm:

Parallel to the RCT, observational data will be collected from a cohort undergoing flexible cystoscopy or intravesical instillation under standard care conditions. This will allow comparison with historical and real-world data, provide additional context for generalizability, and help inform the feasibility of widespread adoption of interventions.

Participant Population Participants will include adults undergoing flexible cystoscopy or bladder instillation for bladder cancer. Eligibility is broad to maximize generalizability, with minimal exclusion criteria. Translation services and literacy supports will be offered to ensure equitable participation.

Study Procedures

* All participants will undergo flexible cystoscopy or intravesical instillation as clinically indicated.
* RCT participants will be randomized to intervention vs. standard care groups.
* Participants will complete short questionnaires before, during, and after the procedure assessing comfort, pain, and anxiety.
* Follow-up will include willingness to undergo repeat procedures and satisfaction ratings.

Outcomes

* Primary outcomes: Patient-reported pain and anxiety scores.
* Secondary outcomes: Overall satisfaction, willingness to repeat procedure, efficiency measures, and clinician feedback.

Significance This study will generate high-quality evidence on practical, low-cost, and easily implementable interventions to improve the patient experience during routine urological procedures. Findings may inform best practice guidelines, enhance patient-centered care, and support broader adoption of comfort-enhancing strategies in cystoscopy services.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of bladder cancer undergoing diagnostic/surveillance flexible cystoscopy or intravesical bladder instillation in the outpatient urology clinic
* Able to provide informed consent

Exclusion Criteria:

Individuals <18 years of age.

* Individuals unable to provide informed consent (e.g., diminished or fluctuating capacity).
* Individuals unable to communicate verbally with study staff (e.g., severe speech/hearing impairment without assistive support available).
* Individuals with severe cognitive impairment or acute distress at the time of approach that prevents informed consent.
* Individuals with known hypersensitivity or allergy to lidocaine, topical anesthetic gel, or any components used in the procedure.
* Individuals for whom, in the opinion of the treating urologist, participation would pose undue clinical risk or interfere with urgent clinical care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Anxiety (VAS 0-100) | Before and immediately after the procedure (within 30 minutes).
  Anxiety level reported by participants immediately following flexible cystoscopy or bladder instillation, measured on a 0-100 visual analogue scale (0 = no anxiety, 100 = worst possible anxiety).
Patient-reported Anxiety (VAS 0-100) | Immediately after the procedure (within 30 minutes).
  Pain/discomfort reported by participants immediately following flexible cystoscopy or bladder instillation, measured on a 0-100 visual analogue scale (0 = no pain, 100 = worst possible pain).

SECONDARY OUTCOMES:
Change in Anxiety from Baseline (VAS 0-100) | Before and immediately after procedure (within 30 minutes).
  Difference in anxiety score from pre-procedure to post-procedure, measured using the 0-100 visual analogue scale.
Baseline Anxiety (GAD-7 Score) | At baseline (pre-procedure, prior to randomization).
  Participant baseline anxiety assessed using the Generalized Anxiety Disorder 7-item (GAD-7) questionnaire. Each item is scored 0-3; total score ranges 0-21, with higher scores indicating greater baseline anxiety.
Patient Satisfaction (Survey-based) | Immediately post-procedure and within 24 hours.
  Patient-reported satisfaction with procedure experience, measured using a structured post-procedure survey (includes overall satisfaction, willingness to repeat, perceived helpfulness of interventions, comparison to expectations, likelihood to recommend, and post-procedure symptoms).
Quality of Life (EORTC QLQ-C30 Global Health Status) | Prior to procedure
  Patient-reported quality of life assessed using the European Organisation for Research and Treatment of Cancer QLQ-C30 questionnaire. Includes global health status and functional scales (0-100).

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital - London Health Sciences Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary results will be made available to researchers upon reasonable request, beginning 12 months after publication. Requests will require a methodologically sound proposal and approval by the study steering committee. Data will be shared via secure transfer after execution of a data use agreement.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting documents will be available beginning 12 months after publication of the primary results, for a period of 5 years.
Access Criteria: De-identified individual participant data (IPD) underlying published results will be made available to qualified researchers upon reasonable request. Access will be limited to investigators with a methodologically sound proposal addressing a scientifically valid research question. Requests must be reviewed and approved by the study steering committee. A data use agreement will be required prior to release. Data and supporting documents (protocol, SAP) will be shared via secure electronic transfer.